CLINICAL TRIAL: NCT02113917
Title: The Formation of a Cohort of HLHa Patients in Order to Study Their Physiopathological Characteristics
Brief Title: Children and Adult Hemophagocytic Syndrome (HLHa)
Acronym: HLH-genes
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Laboratory of normal and pathological development Immune System - IFR 94 U768 (Unknown); Reference Centre for Hereditary Immunodeficiency: CEREDIH (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: NI10015; AOM 10219
Record Dates: First submitted 2013-05-24; First posted 2014-04-15 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Hemophagocytic Syndrome
Keywords: infant, adolescent and adult Hemophagocytic Syndrome; Hemophagocytic lymphohistiocytosis
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood and serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- hemophagocytic syndrome: patient with hemophagocytic syndrome
  Interventions: Biological: Identification of biological markers

INTERVENTIONS:
Biological: Identification of biological markers

SUMMARY:
Different study of HLHa patients :

* Diagnosis criteria, because criteria are based on pediatric genetic studies.
* Physiopathological studies: genetic studies have demonstrated the role of CD8+ cells, in particular because they have a genetic defect affecting their cytotoxic functions in HLH pediatric. the aim is to establish if the same defect is found in both some or in all of HLHa patients. If this is the case, to then establish whether hypomorphic genetic mutations are responsible.

DETAILED DESCRIPTION:
Formation of a prospective and retrospective infant, adolescent and adult HLH patients cohort.

Collection of clinical and biological, therapeutics, informations, in a register, The collection of information is:

* To identify clinical and biological criteria specific to HLHa
* Classify patients into homogeneous groups, based on clinical biological scalability in particular, with regards to their response to treatment
* Identify and analyze the behavioral therapy Creation of a bank of biological samples for use in the study of the pathophysiology of HLHa.

Background:

The hemophagocytic syndrome in infant, adolescent and adults (HLH) is a serious and often lethal condition. The study of literature series HLHa shows that these syndromes frequently develop in immunocompromised patients (renal transplant, HIV, collagen in Processing immunosuppressants) in the course of a viral infection. HLH syndrome has also been described as a clinical form of lymphoma or connective disease (lupus). These clinical forms are rare, severe and recurrent suggesting the possibility that immune deficiency could be involved. The study of pediatric forms has definitely established a link between HLH syndrome and the presence of immune deficiency by identifying the nature of the latter. Four genetically determined diseases are manifested by HLH syndrome. These conditions are Family lymphohistiocytosis (LHF) syndrome, Chediak-Higashi CHS syndrome, Griscelli (GS) type 2 syndromes and X-linked lymphoproliferative (XLP 1 and 2). The mutated genes are respectively perforin Unc 13.4 and syntaxin in the LHF2, 3, 4 (10q locus genetic for LHF 1), CHS1/LYST (Lysosomal Trafficking regulator) in the CHS, in the Rab27a GS type 2, and XIAP and SH2D1A in the XLP. It is now well established that proteins encoded by these genes are necessary for the cytotoxic function of CD8 + and in the absence of these proteins is the cytotoxocity CD8 + deficient. Also, closed clinical and biological characteristics shared by pediatric genetic and adult forms suggest the existence of immune defects responsible for some or all HLH adult patients.

ELIGIBILITY:
Inclusion Criteria:

Major criteria:

* hemophagocytosis found in a specimen histology.
* Fever
* Splenomegaly

Minor criteria:

* adenopathy
* cytopenia> 2 cell lines Hemoglobin <9 g / dl (less than 4 weeks and> 12 g / dl) Platelets <100 000 x 10 / l Neutrophils <1 10 / l
* hypertriglyceridaemia and / or hypofibrinogenaemia Elevated triglycerides> 3 mmol / l Fibrinogen <1.5 g / l
* Ferritin> 500 microg / L

These criteria will be those used for the diagnosis of HLH in adults:

One major criterion and two minor (including hyper ferritin or hypertriglyceridemia) 3 minor criteria (including hyper ferritin or hypertriglyceridemia)

Exclusion Criteria:

* Pregnant women
* A person under guardianship
* Patients under the age of 2 years

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Infant, Adolescent and adult patients who have a HLH syndrome regardless of etiology, hospitalized in Internal Medicine, Critical Care, Hematology, Rheumatology Neurology or Organ Transplantation
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2010-01; Primary Completion 2016-01 (Actual); Study Completion 2017-01-12 (Actual)

PRIMARY OUTCOMES:
biologicals criteria | T0 (before traitment
  measure of : cytokines expression (mmol/L) Hemoglobin (g/dl) number of Platelets (number/L) number of Neutrophils (number/L) number of triglycerides (mmol/L) number of fibrinogen (g/L) number of Ferritin (microg/L)
name of treatment | T2 (T2 is the first day of treatment)
  administrated treatments
Clinicals criteria | T0
  clinicals description of patients : Fever, Splenomegaly and adenopathy
biologicals criteria | T1 (T1 is the first day of HLH syndrome)
  measure of : cytokines expression Hemoglobin level number of Platelets number of Neutrophils number of triglycerides> number of fibrinogen number of Ferritin
biologicals criteria | T2 (T2 is the first day of treatment)
  measure of : cytokines expression Hemoglobin level number of Platelets number of Neutrophils number of triglycerides> number of fibrinogen number of Ferritin
biologicals criteria | T4 (6 /12 months after the resolution of HLH)
  measure of : cytokines expression Hemoglobin level number of Platelets number of Neutrophils number of triglycerides> number of fibrinogen number of Ferritin
Clinicals criteria | T1(T1 is the first day of HLH syndrome)
  clinicals description of patients : Fever, Splenomegaly and adenopathy
Clinicals criteria | T2 (T2 is the first day of treatment)
  clinicals description of patients : Fever, Splenomegaly and adenopathy
Clinicals criteria | T4 6 /12 months after the resolution of HLH)
  clinicals description of patients : Fever, Splenomegaly and adenopathy
name of treatment | T4(6/12 month after resolution of HLH)
  administrated treatments

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Hermine, MD, PhD, Principal Investigator — Hopital Necker Enfants Malades, Assistance Publique des Hôpitaux de Paris
Locations (1):
- Clinical Research Unit, Paris, France

REFERENCES:
- [Derived] Bloch C, Jais JP, Gil M, Boubaya M, Lepelletier Y, Bader-Meunier B, Mahlaoui N, Garcelon N, Lambotte O, Launay D, Larroche C, Lazaro E, Liffermann F, Lortholary O, Michel M, Michot JM, Morel P, Cheminant M, Suarez F, Terriou L, Urbanski G, Viallard JF, Alcais A, Fischer A, de Saint Basile G, Hermine O; French HLH Study Group. Severe adult hemophagocytic lymphohistiocytosis (HLHa) correlates with HLH-related gene variants. J Allergy Clin Immunol. 2024 Jan;153(1):256-264. doi: 10.1016/j.jaci.2023.07.023. Epub 2023 Sep 9. PMID 37678575